CLINICAL TRIAL: NCT04901039
Title: Strategies for Assessment of Fluid Overload in Acute Decompensated Heart Failure
Acronym: FLUID-AHF
Status: Terminated | Type: Observational
Why Stopped: Lack of resources
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-03088
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Decompensated Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Decompensated heart failure: Previously diagnosed heart failure presenting with decompensation to the emergency department
  Interventions: Other: Lung ultrasound; Other: Echocardiography; Other: Peripheral venous pressure; Other: Magnetic resonance imaging; Other: Pulmonary scintigraphy

INTERVENTIONS:
Other: Lung ultrasound — Decompensated HF patients will be evaluated at admission and prior to hospital discharge with a range of tools including lung ultrasound imaging
Other: Echocardiography — Comprehensive echocardiography with evaluation of filling pressures
Other: Peripheral venous pressure — Assessment of peripheral venous pressure
Other: Magnetic resonance imaging — Cardiac magnetic resonance imaging
Other: Pulmonary scintigraphy — Assessment of pulmonary perfusion with scintigraphy

SUMMARY:
Heart failure (HF) is the endstage of all heart disease, characterized by inability of either the left or right heart or both to maintain sufficient output of blood for the demands of the body at normal filling pressures. Patients with HF are often admitted to hospital with decompensation and treated with diuretics. Residual congestion at discharge is associated with increased risk of early rehospitalization and adverse outcomes. However, determination of residual decompensation is complicated and a large number of patients admitted with decompensated heart failure are likely discharged before optimal decongestion has been achieved. Lung ultrasound (LUS) is a promising method to determine residual decompensation with the evaluation of B-lines. In this study our primary aim is to evaluate if LUS together with echocardiographic evaluation of filling pressure according to the European Society of Cardiology (ESC) algorithm performs better than clinical assessment to determine fluid status and risk of early rehospitalization in patients hospitalized for AHF.

ELIGIBILITY:
Inclusion criteria:

Hospitalization for decompensated heart failure is defined as an event that meets all of the following criteria:

1. The patient is admitted to the hospital with a primary diagnosis of HF (previous echo mandatory)
2. The patient's length-of-stay in hospital extends for at least 24 hours
3. The patient exhibits documented new or worsening symptoms due to HF on presentation, including at least ONE of the following:

   * Dyspnea (dyspnea with exertion, dyspnea at rest, orthopnea, paroxysmal nocturnal dyspnea)
   * Decreased exercise tolerance
   * Fatigue
   * Other symptoms of worsened end-organ perfusion or volume overload (as determined by the medical judgement of the investigator)
4. The patient has objective evidence of new or worsening HF, consisting of at least two physical examination findings OR one physical examination finding and at least ONE laboratory criterion, including:

   1. Physical examination findings considered to be due to heart failure, including new or worsened:

      * Peripheral edema
      * Increasing abdominal distention or ascites (in the absence of primary hepatic disease)
      * Pulmonary rales/crackles/crepitations
      * Increased jugular venous pressure and/or hepatojugular reflux
      * S3 gallop
      * Clinically significant or rapid weight gain thought to be related to fluid retention
   2. Laboratory evidence of new or worsening HF, if obtained within 24 hours of presentation, including:

      * Increased B-type natriuretic peptide (BNP)/ N-terminal pro-BNP (NT-proBNP) concentrations consistent with decompensation of heart failure (such as BNP > 500 pg/mL or NT-proBNP > 2,000 pg/mL). In patients with chronically elevated natriuretic peptides, a significant increase should be noted above baseline.
      * Radiological evidence of pulmonary congestion
      * Non-invasive diagnostic evidence of clinically significant elevated left- or right-sided ventricular filling pressure or low cardiac output. For example, echocardiographic criteria could include: E/e' > 15 or D-dominant pulmonary venous inflow pattern.
      * Invasive diagnostic evidence with right heart catheterization showing a pulmonary capillary wedge pressure (pulmonary artery occlusion pressure) ≥ 18 mmHg, central venous pressure ≥ 12 mmHg, or a cardiac index < 2.2 L/min/m2
5. The patient receives initiation or intensification of treatment specifically for HF, including at least one of the following:

   * Augmentation in oral diuretic therapy
   * Intravenous diuretic or vasoactive agent (e.g., inotrope, vasopressor, or vasodilator)
   * Mechanical or surgical intervention, including:

     * Mechanical circulatory support (e.g. intra-aortic balloon pump, ventricular assist device, extracorporeal membrane oxygenation, total artificial heart)
     * Mechanical fluid removal (e.g., ultrafiltration, hemofiltration, dialysis)

Exclusion Criteria:

• Acute coronary syndrome, cardiogenic chock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with decompensated heart failure from 3 hospitals in southern Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Rehospitalization/mortality | 2021-2023
  Rehospitalization or death within 30 days due to decompensated heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Heijl, MD, PhD, Study Director — Cardiology Department, Lund University
Locations (3):
- Sweden (3):
  - Helsingborg General Hospital, Helsingborg
  - Skåne University Hospital, Lund
  - Skåne University Hospital, Malmo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Mebazaa A, Yilmaz MB, Levy P, Ponikowski P, Peacock WF, Laribi S, Ristic AD, Lambrinou E, Masip J, Riley JP, McDonagh T, Mueller C, deFilippi C, Harjola VP, Thiele H, Piepoli MF, Metra M, Maggioni A, McMurray JJ, Dickstein K, Damman K, Seferovic PM, Ruschitzka F, Leite-Moreira AF, Bellou A, Anker SD, Filippatos G. Recommendations on pre-hospital and early hospital management of acute heart failure: a consensus paper from the Heart Failure Association of the European Society of Cardiology, the European Society of Emergency Medicine and the Society of Academic Emergency Medicine--short version. Eur Heart J. 2015 Aug 7;36(30):1958-66. doi: 10.1093/eurheartj/ehv066. Epub 2015 May 21. No abstract available. PMID 25998514
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL. 2013 ACCF/AHA guideline for the management of heart failure: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):1810-52. doi: 10.1161/CIR.0b013e31829e8807. Epub 2013 Jun 5. No abstract available. PMID 23741057
- [Background] Gheorghiade M, Follath F, Ponikowski P, Barsuk JH, Blair JE, Cleland JG, Dickstein K, Drazner MH, Fonarow GC, Jaarsma T, Jondeau G, Sendon JL, Mebazaa A, Metra M, Nieminen M, Pang PS, Seferovic P, Stevenson LW, van Veldhuisen DJ, Zannad F, Anker SD, Rhodes A, McMurray JJ, Filippatos G; European Society of Cardiology; European Society of Intensive Care Medicine. Assessing and grading congestion in acute heart failure: a scientific statement from the acute heart failure committee of the heart failure association of the European Society of Cardiology and endorsed by the European Society of Intensive Care Medicine. Eur J Heart Fail. 2010 May;12(5):423-33. doi: 10.1093/eurjhf/hfq045. Epub 2010 Mar 30. PMID 20354029
- [Background] Gheorghiade M, Konstam MA, Burnett JC Jr, Grinfeld L, Maggioni AP, Swedberg K, Udelson JE, Zannad F, Cook T, Ouyang J, Zimmer C, Orlandi C; Efficacy of Vasopressin Antagonism in Heart Failure Outcome Study With Tolvaptan (EVEREST) Investigators. Short-term clinical effects of tolvaptan, an oral vasopressin antagonist, in patients hospitalized for heart failure: the EVEREST Clinical Status Trials. JAMA. 2007 Mar 28;297(12):1332-43. doi: 10.1001/jama.297.12.1332. Epub 2007 Mar 25. PMID 17384438
- [Background] Price S, Platz E, Cullen L, Tavazzi G, Christ M, Cowie MR, Maisel AS, Masip J, Miro O, McMurray JJ, Peacock WF, Martin-Sanchez FJ, Di Somma S, Bueno H, Zeymer U, Mueller C; Acute Heart Failure Study Group of the European Society of Cardiology Acute Cardiovascular Care Association. Expert consensus document: Echocardiography and lung ultrasonography for the assessment and management of acute heart failure. Nat Rev Cardiol. 2017 Jul;14(7):427-440. doi: 10.1038/nrcardio.2017.56. Epub 2017 Apr 27. PMID 28447662